CLINICAL TRIAL: NCT03422172
Title: An Open Label, Phase 1 Study to Evaluate the PK, Safety, Tolerability and Acceptability of Long Acting Injections of the HIV Integrase Inhibitor, Cabotegravir (CAB; GSK1265744) in HIV Uninfected Chinese Men
Brief Title: A Safety, Tolerability, Acceptability, and Pharmacokinetic (PK) Study of Cabotegravir (CAB) in Healthy Human Immunodeficiency Virus (HIV)-Uninfected Chinese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206898
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: HIV Infections
Keywords: GSK1265744; Pre-Exposure Prophylaxis; Human immunodeficiency virus; Cabotegravir; Pharmacokinetics
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Eligible subjects will receive oral doses of CAB for 4 weeks followed by IM dosing with CAB LA at Week 5, Week 9, Week 17, Week 25 and Week 33.
Masking Description: This will be an open-label study; hence, there will be no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Subjects receiving CAB (Experimental): Eligible subjects will receive oral doses of CAB 30 milligrams (mg) tablets once daily for 4 weeks followed by IM injectable suspension of CAB LA 600 mg at Week 5, Week 9, Week 17, Week 25 and Week 33. There will be an approximately 1-week washout period between the last oral dose and the first injection of CAB at Week 5.
  Interventions: Drug: Oral CAB; Drug: CAB LA

INTERVENTIONS:
Drug: Oral CAB — CAB tablet will be formulated as white to almost white, oval shaped, film coated 30 mg tablets, administered orally once daily. The CAB tablets will be packaged in bottles containing 30 tablets each.
Drug: CAB LA — CAB LA is a sterile white to slightly colored suspension containing 200 mg/mL of CAB as free acid for administration by IM injection in gluteus medius.

SUMMARY:
The pre-exposure prophylaxis (PrEP) is an important component in the overall strategy for prevention of HIV infection. Cabotegravir (CAB) is an integrase strand transfer inhibitor currently in development for treatment and prevention of HIV infection. CAB possesses attributes that allow formulation and delivery as a LA parenteral product. CAB is being developed as both oral and long acting (LA) injectable formulations. This study is designed to evaluate the PK, safety, tolerability, and acceptability of CAB LA in adult HIV uninfected Chinese male subjects at low risk for HIV acquisition. Eligible subjects will receive oral CAB during oral phase of the study followed by CAB LA intramuscular (IM) injection during injection phase of the study. Approximately 60 subjects will be screened, of which, approximately 48 subjects will enter the oral phase and 40 subjects will enter the injection phase of the study. The maximum study duration will be approximately 89 weeks including oral phase, injection phase and follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Subjects are male at birth.
* Subjects who have non-reactive point of care (POC) HIV test and undetectable HIV-1 ribose nucleic acid (RNA) at screening.
* At risk of acquiring HIV, defined as having at least one casual male or female sex partner in the past 24 months.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring at the time of screening.
* Capable of giving written informed consent.
* Agree to appropriate use of contraceptive measures during heterosexual intercourse. All subjects should be counseled on safer sexual practices including the use and benefit/risk of effective barrier methods (example given (e.g.), male condom) to reduce the risk of sexually transmitted infections.
* Willing to undergo all required study procedures.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of the following cardiac diseases: myocardial infarction, congestive heart failure, documented hypertrophic cardiomyopathy, sustained ventricular tachycardia.
* Active skin disease or disorder (that is [i.e.], infection, inflammation, dermatitis, eczema, drug rash, psoriasis, urticaria). Mild cases of localized acne or folliculitis or other mild skin condition may not be exclusionary at the discretion of the Investigator of Record or Medical Monitor.
* Subjects determined by the Investigator to have a high risk of seizures, including subjects with an unstable or poorly controlled seizure disorder. A subject with a prior history of seizure may be considered for enrolment if the Investigator believes the risk of seizure recurrence is low. All cases of prior seizure history should be discussed with the Medical Monitor prior to enrolment.
* Any medical condition, including psychiatric conditions that in the judgment of the investigator would interfere with the subject's ability to complete study procedures.
* Subjects who, in the investigator's judgment, poses a significant suicide risk.
* Use of antiretroviral (ARV) therapy (e.g., for Post exposure prophylaxis [PEP] or PrEP) in the past 30 days.
* Use of high dose aspirin or any other anticoagulant or antiplatelet medication that would interfere with the ability to receive IM injections.
* Assessed by the Investigator of Record or designee as being at "high risk" for HIV infection. This may include one or more of the following: the negative partner in an HIV serodiscordant couple where the HIV infected partner is not suppressed; men who exchange sex for goods or money; men who have engaged in any condomless anal intercourse within the past 6 months; men who have had greater than 5 male or female sexual partners within the past 6 months; men who have had a sexually transmitted disease within the past 6 months; any other behavior assessed by the investigator as "high risk".
* History of drug or alcohol consumption that in the opinion of the Principal Investigator will interfere with study participation.
* Ongoing intravenous drug use - episodic use or any use in the past 90 days is exclusionary (as assessed by the study investigator).
* One or more reactive HIV test results at screening or enrolment, even if HIV infection is not confirmed. Negative HIV RNA must also be documented at screening.
* Co-enrolment in any other HIV interventional research study (provided by self-report or other available documentation) or prior enrolment and receipt of the active arm (i.e., NOT a placebo) of a HIV vaccine trial (provided by available documentation).
* Any of the following laboratory values during the screening period: positive hepatitis C antibody result; positive Hepatitis B surface antigen (HBsAg); hemoglobin <11 grams per deciliter (g/dL); absolute neutrophil count <750 cells/ cubic millimeter (mm^3); platelet count <=100,000 cells/mm^3; presence of a coagulopathy as defined by an international normalized ratio(INR)>1.5 or a partial thromboplastin time (PTT) >45 seconds; calculated creatinine clearance <60 milliliter/minute (mL/minute) using the Cockcroft-Gault equation; a single repeat test is allowed during the screening period to verify a result, with the exception of HIV tests.
* Subjects with an ALT, alkaline phosphatase or bilirubin >=1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* The subject has a tattoo or other dermatological condition overlying the gluteus region which may interfere with interpretation of injection site reactions.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy male subjects at low risk of HIV infection will be eligible to participate in this study.
Enrollment: 48 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (3):
- China (3):
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Han K, Wannamaker P, Lu H, Zhu B, Wang M, Paff M, Spreen WR, Ford SL. Safety, Tolerability, Pharmacokinetics, and Acceptability of Oral and Long-Acting Cabotegravir in HIV-Negative Chinese Men. Antimicrob Agents Chemother. 2022 Mar 15;66(3):e0205721. doi: 10.1128/AAC.02057-21. Epub 2022 Feb 7. PMID 35129374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, multi-site study to evaluate pharmacokinetic (PK), safety, tolerability, and acceptability of long acting (LA) injections of cabotegravir (CAB) in human immunodeficieny virus (HIV) uninfected Chinese men.
Pre-assignment Details: A total of 48 participants were enrolled and randomized to receive study treatment. The study consisted of oral lead-in phase (4 weeks), injection phase (weeks 5 to 41) and long-term follow-up phase (weeks 42 to 89).
Groups:
- Cabotegravir: Participants received 30 milligrams (mg) Cabotegravir tablet once daily orally for 4 weeks. Participants who completed the oral lead-in phase, received CAB LA 600 mg administered as a single 3 milliliter (mL) intramuscular (IM) injection on Weeks 5, 9, 17, 25 and 33 during injection phase. There was a washout of 7 days between oral and Injection phase. Participants were followed-up till Week 89 (long-term follow-up phase).
Period: Oral lead-in Phase (4 Weeks)
Arm/Group | Cabotegravir
Started | 48
Completed | 47
Not Completed | 1
Not completed — Adverse Event | 1
Period: Washout (7 Days)
Arm/Group | Cabotegravir
Started | 47
Completed | 47
Not Completed | 0
Period: Injection Phase (Week 5 to Week 41)
Arm/Group | Cabotegravir
Started | 47
Completed | 43
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3
Period: Long Term Follow-up Phase(Upto Week 89)
Arm/Group | Cabotegravir
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cabotegravir
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.1 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious Adverse Events (AEs) and Serious AEs (SAEs): Injection Phase
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, or other situations as per investigator's judgement.
Time Frame: Week 5 to 41
Population: Safety Injection Population. It comprised of all participants who received at least one CAB LA injection.
Measure: Count of Participants; unit: Participants
Groups:
- CAB LA 600 mg (Injection Phase): Participants received CAB LA 600 mg administered as a single 3 mL intramuscular injection on Weeks 5, 9, 17, 25 and 33 during Injection phase.
Arm/Group | CAB LA 600 mg (Injection Phase)
Number analyzed (Participants) | 47
Participants
  Non-serious AEs | 47
  SAEs | 1

2. Primary Outcome: Number of Participants With Maximum Toxicity Post-Baseline in Hematology Parameters-Injection Phase
Description: Hematology parameters were graded according to Division of Acquired Immunodeficiency Syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events as Grade 0: none, Grade 1: mild; Grade 2: moderate; Grade 3: severe; and Grade 4: potentially life-threatening consequences. Higher grade indicates more severity. Clinical hematology parameters included: Activated partial thromboplastin time (APTT) prolonged, hemoglobin (Hb) (increased), white blood cells (WBC) (decreased), lymphocytes count (decreased), neutrophils (decreased), platelets (decreased), prothrombin international normalized ratio (Pro.INR) (increased). Baseline was the last available assessment prior to the time of the first dose. Maximum toxicity grade reached by a participant post-Baseline was summarized.
Time Frame: Week 5 to 41
Population: Safety Injection Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category title).
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg (Injection Phase)
Number analyzed (Participants) | 47
Participants
  APTT prolonged, Grade 0, n=28: number analyzed (Participants) | 28
  APTT prolonged, Grade 0, n=28 | 28
  APTT prolonged, Grade 1, n=28: number analyzed (Participants) | 28
  APTT prolonged, Grade 1, n=28 | 0
  APTT prolonged, Grade 2, n=28: number analyzed (Participants) | 28
  APTT prolonged, Grade 2, n=28 | 0
  APTT prolonged, Grade 3, n=28: number analyzed (Participants) | 28
  APTT prolonged, Grade 3, n=28 | 0
  APTT prolonged, Grade 4, n=28: number analyzed (Participants) | 28
  APTT prolonged, Grade 4, n=28 | 0
  Hb (increased), Grade 0, n=47 | 47
  Hb (increased), Grade 1, n=47 | 0
  Hb (increased), Grade 2, n=47 | 0
  Hb (increased), Grade 3, n=47 | 0
  Hb (increased), Grade 4, n=47 | 0
  WBC (decreased), Grade 0, n=47 | 47
  WBC (decreased), Grade 1, n=47 | 0
  WBC (decreased), Grade 2, n=47 | 0
  WBC (decreased), Grade 3, n=47 | 0
  WBC (decreased), Grade 4, n=47 | 0
  Lymphocytes count (decreased), Grade 0, n=47 | 47
  Lymphocytes count (decreased), Grade 1, n=47 | 0
  Lymphocytes count (decreased), Grade 2, n=47 | 0
  Lymphocytes count (decreased), Grade 3, n=47 | 0
  Lymphocytes count (decreased), Grade 4, n=47 | 0
  Neutrophils (decreased), Grade 0, n=47 | 47
  Neutrophils (decreased), Grade 1, n=47 | 0
  Neutrophils (decreased), Grade 2, n=47 | 0
  Neutrophils (decreased), Grade 3, n=47 | 0
  Neutrophils (decreased), Grade 4, n=47 | 0
  Platelets (decreased), Grade 0, n=47 | 45
  Platelets (decreased), Grade 1, n=47 | 2
  Platelets (decreased), Grade 2, n=47 | 0
  Platelets (decreased), Grade 3, n=47 | 0
  Platelets (decreased), Grade 4, n=47 | 0
  Prothrombin INR (increased), Grade 0, n=28: number analyzed (Participants) | 28
  Prothrombin INR (increased), Grade 0, n=28 | 28
  Prothrombin INR (increased), Grade 1, n=28: number analyzed (Participants) | 28
  Prothrombin INR (increased), Grade 1, n=28 | 0
  Prothrombin INR (increased), Grade 2, n=28: number analyzed (Participants) | 28
  Prothrombin INR (increased), Grade 2, n=28 | 0
  Prothrombin INR (increased),Grade 3, n=28: number analyzed (Participants) | 28
  Prothrombin INR (increased),Grade 3, n=28 | 0
  Prothrombin INR (increased), Grade 4, n=28: number analyzed (Participants) | 28
  Prothrombin INR (increased), Grade 4, n=28 | 0

3. Primary Outcome: Number of Participants With Maximum Toxicity Post-Baseline in Chemistry Parameters: Injection Phase
Description: Chemistry parameters were graded according to DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events as Grade 0: none, Grade 1: mild; Grade 2: moderate; Grade 3: severe; and Grade 4: potentially life-threatening consequences. Higher grade indicates more severity. Clinical chemistry laboratory parameters included alanine amino transferase (ALT), albumin, alkaline phosphatase (ALP), Aspartate Aminotransferase (AST), bilirubin, calcium (hypercalcemia and hypocalcemia), carbon dioxide (CO2) (decreased), cholesterol (high), Creatine phosphokinase (CPK) increased, Creatinine increased, creatinine clearance (decreased), glucose (hyperglycemia and hypoglycemia), Hypophosphatemia, Potassium (Hyperkalemia and hypokalemia), Sodium (hypernatremia and hyponatremia), Hypertriglyceridemia, uric acid (increased). Baseline was the last available assessment prior to the time of the first dose. Maximum toxicity grade reached by a participant post-Baseline was summarized.
Time Frame: Week 5 to 41
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg (Injection Phase)
Number analyzed (Participants) | 47
Participants
  ALT, Grade 0, n=47 | 41
  ALT, Grade 1, n=47 | 6
  ALT, Grade 2, n=47 | 0
  ALT, Grade 3, n=47 | 0
  ALT, Grade 4, n=47 | 0
  Albumin, Grade 0, n=47 | 47
  Albumin, Grade 1, n=47 | 0
  Albumin, Grade 2, n=47 | 0
  Albumin, Grade 3, n=47 | 0
  Albumin, Grade 4, n=47 | 0
  ALP, Grade 0, n=47 | 47
  ALP, Grade 1, n=47 | 0
  ALP, Grade 2, n=47 | 0
  ALP, Grade 3, n=47 | 0
  ALP, Grade 4, n=47 | 0
  AST, Grade 0, n=47 | 39
  AST, Grade 1, n=47 | 6
  AST, Grade 2, n=47 | 2
  AST, Grade 3, n=47 | 0
  AST, Grade 4, n=47 | 0
  Bilirubin, Grade 0, n=47 | 45
  Bilirubin, Grade 1, n=47 | 2
  Bilirubin, Grade 2, n=47 | 0
  Bilirubin, Grade 3, n=47 | 0
  Bilirubin, Grade 4, n=47 | 0
  Calcium, Hypercalcemia, Grade 0, n=47 | 47
  Calcium, Hypercalcemia, Grade 1, n=47 | 0
  Calcium, Hypercalcemia, Grade 2, n=47 | 0
  Calcium, Hypercalcemia, Grade 3, n=47 | 0
  Calcium, Hypercalcemia, Grade 4, n=47 | 0
  Calcium, Hypocalcemia, Grade 0, n=47 | 47
  Calcium, Hypocalcemia, Grade 1, n=47 | 0
  Calcium, Hypocalcemia, Grade 2, n=47 | 0
  Calcium, Hypocalcemia, Grade 3, n=47 | 0
  Calcium, Hypocalcemia, Grade 4, n=47 | 0
  CO2 decreased, Grade 0, n=47 | 47
  CO2 decreased, Grade 1, n=47 | 0
  CO2 decreased, Grade 2, n=47 | 0
  CO2 decreased Grade 3, n=47 | 0
  CO2 decreased, Grade 4, n=47 | 0
  Cholesterol (High), Grade 0, n=28: number analyzed (Participants) | 28
  Cholesterol (High), Grade 0, n=28 | 26
  Cholesterol (High), Grade 1, n=28: number analyzed (Participants) | 28
  Cholesterol (High), Grade 1, n=28 | 2
  Cholesterol (High), Grade 2, n=28: number analyzed (Participants) | 28
  Cholesterol (High), Grade 2, n=28 | 0
  Cholesterol (High), Grade 3, n=28: number analyzed (Participants) | 28
  Cholesterol (High), Grade 3, n=28 | 0
  Cholesterol (High), Grade 4, n=28: number analyzed (Participants) | 28
  Cholesterol (High), Grade 4, n=28 | 0
  CPK increased, Grade 0, n=47 | 38
  CPK increased, Grade 1, n=47 | 4
  CPK increased, Grade 2, n=47 | 0
  CPK increased, Grade 3, n=47 | 4
  CPK increased, Grade 4, n=47 | 1
  Creatinine increased, Grade 0, n=47 | 46
  Creatinine increased, Grade 1, n=47 | 1
  Creatinine increased, Grade 2, n=47 | 0
  Creatinine increased, Grade 3, n=47 | 0
  Creatinine increased, Grade 4, n=47 | 0
  Creatinine clearance decreased, Grade 0, n=47 | 31
  Creatinine clearance decreased, Grade 1, n=47 | 0
  Creatinine clearance decreased, Grade 2, n=47 | 16
  Creatinine clearance decreased, Grade 3, n=47 | 0
  Creatinine clearance decreased, Grade 4, n=47 | 0
  Glucose (hyperglycemia), Grade 0, n=47 | 38
  Glucose (hyperglycemia), Grade 1, n=47 | 7
  Glucose (hyperglycemia), Grade 2, n=47 | 2
  Glucose (hyperglycemia), Grade 3, n=47 | 0
  Glucose (hyperglycemia), Grade 4, n=47 | 0
  Glucose (hypoglycemia), Grade 0, n=47 | 46
  Glucose (hypoglycemia), Grade 1, n=47 | 1
  Glucose (hypoglycemia), Grade 2, n=47 | 0
  Glucose (hypoglycemia), Grade 3, n=47 | 0
  Glucose (hypoglycemia), Grade 4, n=47 | 0
  Hypophosphatemia, Grade 0, n=47 | 45
  Hypophosphatemia, Grade 1, n=47 | 2
  Hypophosphatemia, Grade 2, n=47 | 0
  Hypophosphatemia, Grade 3, n=47 | 0
  Hypophosphatemia, Grade 4, n=47 | 0
  Potassium (Hyperkalemia), Grade 0, n=47 | 47
  Potassium (Hyperkalemia), Grade 1, n=47 | 0
  Potassium (Hyperkalemia), Grade 2, n=47 | 0
  Potassium (Hyperkalemia), Grade 3, n=47 | 0
  Potassium (Hyperkalemia), Grade 4, n=47 | 0
  Potassium (Hypokalemia), Grade 0, n=47 | 47
  Potassium (Hypokalemia), Grade 1, n=47 | 0
  Potassium (Hypokalemia), Grade 2, n=47 | 0
  Potassium (Hypokalemia), Grade 3, n=47 | 0
  Potassium (Hypokalemia), Grade 4, n=47 | 0
  Sodium, hypernatremia, Grade 0, n=47 | 47
  Sodium, hypernatremia, Grade 1, n=47 | 0
  Sodium, hypernatremia, Grade 2, n=47 | 0
  Sodium, hypernatremia, Grade 3, n=47 | 0
  Sodium, hypernatremia, Grade 4, n=47 | 0
  Sodium, hyponatremia, Grade 0, n=47 | 47
  Sodium, hyponatremia, Grade 1, n=47 | 0
  Sodium, hyponatremia, Grade 2, n=47 | 0
  Sodium, hyponatremia, Grade 3, n=47 | 0
  Sodium, hyponatremia, Grade 4, n=47 | 0
  Hypertriglyceridemia, Grade 0, n=28: number analyzed (Participants) | 28
  Hypertriglyceridemia, Grade 0, n=28 | 21
  Hypertriglyceridemia, Grade 1, n=28: number analyzed (Participants) | 28
  Hypertriglyceridemia, Grade 1, n=28 | 6
  Hypertriglyceridemia, Grade 2, n=28: number analyzed (Participants) | 28
  Hypertriglyceridemia, Grade 2, n=28 | 1
  Hypertriglyceridemia, Grade 3, n=28: number analyzed (Participants) | 28
  Hypertriglyceridemia, Grade 3, n=28 | 0
  Hypertriglyceridemia, Grade 4, n=28: number analyzed (Participants) | 28
  Hypertriglyceridemia, Grade 4, n=28 | 0
  Uric acid increased, Grade 0, n=47 | 32
  Uric acid increased, Grade 1, n=47 | 14
  Uric acid increased, Grade 2, n=47 | 1
  Uric acid increased ,Grade 3, n=47 | 0
  Uric acid increased, Grade 4, n=47 | 0

4. Primary Outcome: Number of Participants With Maximum Toxicity Post-Baseline in Urinalysis Parameters: Injection Phase
Description: Urinalysis parameters were graded according to DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events as Grade 0: none, Grade 1: mild; Grade 2: moderate; Grade 3: severe; and Grade 4: potentially life-threatening consequences. Urinalysis parameters included: Protein. Baseline was the last available assessment prior to the time of the first dose. Maximum toxicity grade reached by a participant post-Baseline was summarized.
Time Frame: Week 5 to 41
Population: Safety Injection Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg (Injection Phase)
Number analyzed (Participants) | 29
Participants
  Protein, Grade 0 | 29
  Protein, Grade 1 | 0
  Protein, Grade 2 | 0
  Protein, Grade 3 | 0
  Protein, Grade 4 | 0

5. Primary Outcome: Number of Participants With Shift From Baseline in Vital Signs With Respect to Clinical Concern Range: Injection Phase
Description: Vital signs were measured after participants had rested in supine position for at least 5 minutes. Clinical concern ranges were: systolic blood pressure (SBP) (Low: <85 millimeters of mercury [mmHg], High: >160 mmHg), diastolic blood pressure (DBP) (Low: <45 mmHg, High: >100 mmHg), pulse rate (Low: <40 mmHg, High: >100 mmHg). Worst case results are presented. Participants were counted in the worst case category that their value changes to (Low, Normal or High), unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, were recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Time Frame: Week 5 to 41
Population: Safety Injection Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg (Injection Phase)
Number analyzed (Participants) | 47
Participants
  SBP, To low | 0
  SBP, To Normal or No Change | 46
  SBP, To High | 1
  DBP, To low | 0
  DBP, To Normal or No Change | 46
  DBP, To High | 1
  Pulse rate, To low | 0
  Pulse rate, To Normal or No Change | 46
  Pulse rate, To High | 1

6. Primary Outcome: Number of Participants Withdrawn Due to AEs- Injection Phase
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Number of participants withdrawn from study due to AEs is presented.
Time Frame: Week 5 to 41
Population: Safety Injection Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg (Injection Phase)
Number analyzed (Participants) | 47
Participants | 0

7. Primary Outcome: Number of Participants Experiencing Injection Site Reactions (ISR)-Injection Phase
Description: Injection site reactions were recorded via ISR diaries and managed through investigator assessment. Number of participants who experienced any injection site reaction (like pain, itching, bruising, bump, discoloration, redness, skin firmness, swelling, warm to touch etc.) is presented.
Time Frame: Week 5 to 41
Population: Safety Injection Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg (Injection Phase)
Number analyzed (Participants) | 47
Participants | 47

8. Primary Outcome: Concentration of Cabotegravir in Plasma at the End of the Dosing Interval (Ctau)-Oral lead-in Phase
Description: Blood samples were collected at the indicated time points for the determination of Ctau following oral dose of Cabotegravir and was calculated by standard non-compartmental analysis.
Time Frame: Day 27: Pre-dose and at 1, 2, 3, 4, 8, 24 and 168 hours post-dose
Population: Oral Pharmacokinetic (PK) Population. It consisted of all participants in the 'Safety Population' for whom an intensive oral PK sample was obtained and analyzed. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Groups:
- CAB 30 mg (Oral lead-in Phase): Participants received 30 mg Cabotegravir tablet once daily orally for 4 weeks during oral lead-in phase.
Arm/Group | CAB 30 mg (Oral lead-in Phase)
Number analyzed (Participants) | 17
Micrograms per milliliter | 6.807 (26.8)

9. Primary Outcome: Area Under the Plasma Concentration Time Curve Over the Dosing Interval (AUC[0-tau]) Following Oral Dosing of Cabotegravir-Oral lead-in Phase
Description: Blood samples were collected at the indicated time points for the determination of AUC(0-tau) following oral dose of Cabotegravir and was calculated by standard non-compartmental analysis.
Time Frame: Day 27: Pre-dose and at 1, 2, 3, 4, 8, 24 and 168 hours post-dose
Population: Oral PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter
Arm/Group | CAB 30 mg (Oral lead-in Phase)
Number analyzed (Participants) | 17
Hour*micrograms per milliliter | 191.1 (20.5)

10. Primary Outcome: Maximum Observed Concentration (Cmax) Following Oral Dosing With Cabogegravir-Oral lead-in Phase
Description: Blood samples were collected at the indicated time points for the determination of Cmax following oral dose of Cabotegravir and was calculated by standard non-compartmental analysis.
Time Frame: Day 27: Pre-dose and at 1, 2, 3, 4, 8, 24 and 168 hours post-dose
Population: Oral PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | CAB 30 mg (Oral lead-in Phase)
Number analyzed (Participants) | 17
Micrograms per milliliter | 10.447 (19.5)

11. Primary Outcome: Time of Occurrence of Cmax (Tmax) Following Oral Dosing With Cabotegravir-Oral lead-in Phase
Description: Blood samples were collected at the indicated time points for the determination of Tmax following oral dose of Cabotegravir and was calculated by standard non-compartmental analysis.
Time Frame: Day 27: Pre-dose and at 1, 2, 3, 4, 8, 24 and 168 hours post-dose
Population: Oral PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | CAB 30 mg (Oral lead-in Phase)
Number analyzed (Participants) | 17
Hours | 2.0000 [0.983 to 4.000]

12. Primary Outcome: Apparent Clearance Following Oral Dosing (CL/F) Following Dosing With Cabotegravir-Oral lead-in Phase
Description: Blood samples were collected at the indicated time points for the determination of CL/F following oral dose of Cabotegravir and was calculated by standard non-compartmental analysis.
Time Frame: Day 27: Pre-dose and at 1, 2, 3, 4, 8, 24 and 168 hours post-dose
Population: Oral PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | CAB 30 mg (Oral lead-in Phase)
Number analyzed (Participants) | 17
Liters per hour | 0.1570 (20.5)

13. Primary Outcome: Terminal Absorption Elimination Half-life (t1/2) Following Oral Dosing With Cabotegravir-Oral lead-in Phase
Description: Blood samples were collected at the indicated time points for the determination of t1/2 following oral dose of Cabotegravir and was calculated by standard non-compartmental analysis.
Time Frame: Day 27: Pre-dose and at 1, 2, 3, 4, 8, 24 and 168 hours post-dose
Population: Oral PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | CAB 30 mg (Oral lead-in Phase)
Number analyzed (Participants) | 17
Hours | 45.24 (20.5)

14. Primary Outcome: Apparent Terminal Phase Rate Constant (Lambda z) Following Oral Dosing With Cabotegravir-Oral lead-in Phase
Description: Blood samples were collected at the indicated time points for the determination of Lambda z following oral dose of Cabotegravir and was calculated by standard non-compartmental analysis.
Time Frame: Day 27: Pre-dose and at 1, 2, 3, 4, 8, 24 and 168 hours post-dose
Population: Oral PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | CAB 30 mg (Oral lead-in Phase)
Number analyzed (Participants) | 17
Per hour | 0.01532 (20.5)

15. Primary Outcome: Volume of Distribution at Steady State (Vss) Following Oral Dosing With Cabotegravir-Oral lead-in Phase
Description: Blood samples were collected at the indicated time points for the determination of Vss following oral dose of Cabotegravir and was calculated by standard non-compartmental analysis.
Time Frame: Day 27: Pre-dose and at 1, 2, 3, 4, 8, 24 and 168 hours post-dose
Population: Oral PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | CAB 30 mg (Oral lead-in Phase)
Number analyzed (Participants) | 17
Liters | 10.246 (17.8)

16. Primary Outcome: Ctau Following IM Dosing With CAB LA During Injection Phase
Description: Blood samples were collected at the indicated time points for the determination of Ctau following IM dose of CAB LA and was calculated by standard non-compartmental analysis.
Time Frame: Pre-dose sample on Weeks 5, 9, 17, 25, 33; Post-dose sample on Weeks 6, 10, 18, 26, 34, 37, 41
Population: Injection (Week 41) PK Population. It consisted of all participants in the 'Safety Population' for whom an injection PK sample was obtained and analyzed during Weeks 5 to 41. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | CAB LA 600 mg (Injection Phase)
Number analyzed (Participants) | 43
Micrograms per milliliter | 1.5831 (43.1)

17. Primary Outcome: AUC(0-tau) Following IM Dosing With CAB LA During Injection Phase
Description: Blood samples were collected at the indicated time points for the determination of AUC (0-tau) following IM dose of CAB LA and was calculated by standard non-compartmental analysis.
Time Frame: Pre-dose sample on Weeks 5, 9, 17, 25, 33; Post-dose sample on Weeks 6, 10, 18, 26, 34, 37, 41
Population: Injection (Week 41) PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter
Arm/Group | CAB LA 600 mg (Injection Phase)
Number analyzed (Participants) | 43
Hour*micrograms per milliliter | 3415.1 (41.9)

18. Primary Outcome: Cmax Following IM Dosing With CAB LA During Injection Phase
Description: Blood samples were collected at the indicated time points for the determination of Cmax following IM dose of CAB LA and was calculated by standard non-compartmental analysis.
Time Frame: Pre-dose sample on Weeks 5, 9, 17, 25, 33; Post-dose sample on Weeks 6, 10, 18, 26, 34, 37, 41
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | CAB LA 600 mg (Injection Phase)
Number analyzed (Participants) | 44
Micrograms per milliliter | 3.730 (66.1)

19. Primary Outcome: Tmax Following IM Dosing With CAB LA During Injection Phase
Description: Blood samples were collected at the indicated time points for the determination of Tmax following IM dose of CAB LA and was calculated by standard non-compartmental analysis.
Time Frame: Pre-dose sample on Weeks 5, 9, 17, 25, 33; Post-dose sample on Weeks 6, 10, 18, 26, 34, 37, 41
Population: as for outcome 17
Measure: Median (Full Range); unit: Hour
Arm/Group | CAB LA 600 mg (Injection Phase)
Number analyzed (Participants) | 44
Hour | 167.433 [0.00 to 765.25]

20. Secondary Outcome: Ctau Following IM Dosing With CAB LA Through Injection and Long-term Follow-up Phases
Description: as for outcome 16
Time Frame: Pre-dose sample on Weeks 5, 9, 17, 25, 33; Post-dose sample on Weeks 6, 10, 18, 26, 34, 37, 41, 53, 65, 77, 89
Population: Injection (Week 89) PK Population. It consisted of all participants in the 'Safety Population' for whom an injection PK sample was obtained and analyzed during Weeks 5 to 89 (through Injection and long-term follow-up phases). Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Groups:
- CAB LA 600 mg (Injection Phase and Long-term Follow up): Participants received CAB LA 600 mg administered as a single 3 mL intramuscular injection on Weeks 5, 9, 17, 25 and 33 during Injection phase followed by a long term follow up from Week 41 to 89.
Arm/Group | CAB LA 600 mg (Injection Phase and Long-term Follow up)
Number analyzed (Participants) | 43
Micrograms per milliliter | 1.5831 (43.1)

21. Secondary Outcome: AUC(0-tau) Following IM Dosing With CAB LA Through Injection and Long-term Follow-up Phases
Description: Blood samples were collected at the indicated time points for the determination of AUC(0-tau) following IM dose of CAB LA and was calculated by standard non-compartmental analysis.
Time Frame: Pre-dose sample on Weeks 5, 9, 17, 25, 33; Post-dose sample on Weeks 6, 10, 18, 26, 34, 37, 41, 53, 65, 77, 89
Population: Injection (Week 89) PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter
Arm/Group | CAB LA 600 mg (Injection Phase and Long-term Follow up)
Number analyzed (Participants) | 43
Hour*micrograms per milliliter | 3442.5 (41.1)

22. Secondary Outcome: Cmax Following IM Dosing With CAB LA Through Injection and Long-term Follow-up Phases
Description: as for outcome 18
Time Frame: Pre-dose sample on Weeks 5, 9, 17, 25, 33; Post-dose sample on Weeks 6, 10, 18, 26, 34, 37, 41, 53, 65, 77, 89
Population: Injection (Week 89) (PK) Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | CAB LA 600 mg (Injection Phase and Long-term Follow up)
Number analyzed (Participants) | 44
Micrograms per milliliter | 3.730 (66.1)

23. Secondary Outcome: Tmax Following IM Dosing With CAB LA Through Injection and Long-term Follow-up Phases
Description: as for outcome 19
Time Frame: Pre-dose sample on Weeks 7 9, 17, 25, 33; Post-dose sample on Weeks 6, 10, 18, 26, 34, 37, 41, 53, 65, 77, 89
Population: as for outcome 21
Measure: Median (Full Range); unit: Hour
Arm/Group | CAB LA 600 mg (Injection Phase and Long-term Follow up)
Number analyzed (Participants) | 44
Hour | 167.433 [0.00 to 765.25]

24. Secondary Outcome: CL/F Following IM Dosing With CAB LA Through Injection and Long-term Follow-up Phases
Description: Blood samples were collected at the indicated time points for the determination of CL/F following IM dose of CAB LA and was calculated by standard non-compartmental analysis.
Time Frame: Pre-dose sample on Weeks 7, 9, 17, 25, 33; Post-dose sample on Weeks 6, 10, 18, 26, 34, 37, 41, 53, 65, 77, 89
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | CAB LA 600 mg (Injection Phase and Long-term Follow up)
Number analyzed (Participants) | 43
Liters per hour | 0.17429 (41.1)

25. Secondary Outcome: T1/2 Following IM Dosing With CAB LA Through Injection and Long-term Follow-up Phases
Description: Blood samples were collected at the indicated time points for the determination of t1/2 following IM dose of CAB LA and was calculated by standard non-compartmental analysis.
Time Frame: Pre-dose sample on Weeks 5, 9, 17, 25, 33; Post-dose sample on Weeks 6, 10, 18, 26, 34, 37, 41, 53, 65, 77, 89
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | CAB LA 600 mg (Injection Phase and Long-term Follow up)
Number analyzed (Participants) | 41
Hour | 1128.6 (71.2)

26. Secondary Outcome: Lambda z Following IM Dosing With CAB LA Through Injection and Long-term Follow-up Phases
Description: Blood samples were collected at the indicated time points for the determination of Lambda z following IM dose of CAB LA and was calculated by standard non-compartmental analysis.
Time Frame: Pre-dose sample on Weeks 5, 9, 17, 25, 33; Post-dose sample on Weeks 6, 10, 18, 26, 34, 37, 41, 53, 65, 77, 89
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | CAB LA 600 mg (Injection Phase and Long-term Follow up)
Number analyzed (Participants) | 41
Per hour | 0.0006141 (71.2)

27. Secondary Outcome: Vss Following IM Dosing With CAB LA Through Injection and Long-term Follow-up Phases
Description: Blood samples were collected at the indicated time points for the determination of Vss following IM dose of CAB LA and was calculated by standard non-compartmental analysis.
Time Frame: Pre-dose sample on Weeks 5, 9, 17, 25, 33; Post-dose sample on Weeks 6, 10, 18, 26, 34, 37, 41, 53, 65, 77, 89
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | CAB LA 600 mg (Injection Phase and Long-term Follow up)
Number analyzed (Participants) | 41
Liters | 282.44 (124.8)

28. Secondary Outcome: Number of Participants With Non-serious AEs and SAEs (Oral lead-in Phase)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose results in death, Is life-threatening, Requires inpatient hospitalization or prolongation of existing hospitalization, Results in persistent disability/incapacity, Is a congenital anomaly/birth defect, other situation as per investigator's judgement.
Time Frame: Up to Week 4
Population: Safety Population. It comprised all participants who received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB 30 mg (Oral lead-in Phase)
Number analyzed (Participants) | 48
Participants
  Non-serious AEs | 13
  SAEs | 0

29. Secondary Outcome: Number of Participants Withdrawn Due to AEs-oral lead-in Phase
Description: as for outcome 6
Time Frame: Up to Week 4
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB 30 mg (Oral lead-in Phase)
Number analyzed (Participants) | 48
Participants | 1

30. Secondary Outcome: Number of Participants With Maximum Toxicity Post-Baseline in Chemistry Parameters: Oral lead-in Phase
Description: Chemistry parameters were graded according to DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events as Grade 0: none, Grade 1: mild; Grade 2: moderate; Grade 3: severe; and Grade 4: potentially life-threatening consequences. Higher grade indicates more severity. Clinical chemistry laboratory parameters included ALT, albumin, ALP, AST, bilirubin, calcium (hypercalcemia and hypocalcemia), CO2 decreased, cholesterol, CPK increased, Creatinine increased, creatinine clearance (decreased), glucose (hyperglycemia and hypoglycemia), Hypophosphatemia, Potassium (Hyperkalemia and hypokalemia), Sodium (hypernatremia and hyponatremia), Hypertriglyceridemia, uric acid (increased). Baseline was the last available assessment prior to the time of the first dose. Maximum toxicity grade reached by a participant post-Baseline was summarized.
Time Frame: Up to Week 4
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category title).
Measure: Count of Participants; unit: Participants
Arm/Group | CAB 30 mg (Oral lead-in Phase)
Number analyzed (Participants) | 48
Participants
  ALT, Grade 0, n=48 | 45
  ALT, Grade 1, n=48 | 3
  ALT, Grade 2, n=48 | 0
  ALT, Grade 3, n=48 | 0
  ALT, Grade 4, n=48 | 0
  Albumin, Grade 0, n=48 | 48
  Albumin, Grade 1, n=48 | 0
  Albumin, Grade 2, n=48 | 0
  Albumin, Grade 3, n=48 | 0
  Albumin, Grade 4, n=48 | 0
  ALP, Grade 0, n=48 | 48
  ALP, Grade 1, n=48 | 0
  ALP, Grade 2, n=48 | 0
  ALP, Grade 3, n=48 | 0
  ALP, Grade 4, n=48 | 0
  AST, Grade 0, n=48 | 47
  AST, Grade 1, n=48 | 1
  AST, Grade 2, n=48 | 0
  AST, Grade 3, n=48 | 0
  AST, Grade 4, n=48 | 0
  Bilirubin, Grade 0, n=48 | 48
  Bilirubin, Grade 1, n=48 | 0
  Bilirubin, Grade 2, n=48 | 0
  Bilirubin, Grade 3, n=48 | 0
  Bilirubin, Grade 4, n=48 | 0
  Calcium, Hypercalcemia, Grade 0, n=48 | 48
  Calcium, Hypercalcemia, Grade 1, n=48 | 0
  Calcium, Hypercalcemia, Grade 2, n=48 | 0
  Calcium, Hypercalcemia, Grade 3, n=48 | 0
  Calcium, Hypercalcemia, Grade 4, n=48 | 0
  Calcium, Hypocalcemia, Grade 0, n=48 | 48
  Calcium, Hypocalcemia, Grade 1, n=48 | 0
  Calcium, Hypocalcemia, Grade 2, n=48 | 0
  Calcium, Hypocalcemia, Grade 3, n=48 | 0
  Calcium, Hypocalcemia, Grade 4, n=48 | 0
  CO2 decreased, Grade 0, n=48 | 47
  CO2 decreased, Grade 1, n=48 | 1
  CO2 decreased, Grade 2, n=48 | 0
  CO2 decreased, Grade 3, n=48 | 0
  CO2 decreased, Grade 4, n=48 | 0
  Cholesterol (High), Grade 0, n=3: number analyzed (Participants) | 3
  Cholesterol (High), Grade 0, n=3 | 3
  Cholesterol (High), Grade 1, n=3: number analyzed (Participants) | 3
  Cholesterol (High), Grade 1, n=3 | 0
  Cholesterol (High), Grade 2, n=3: number analyzed (Participants) | 3
  Cholesterol (High), Grade 2, n=3 | 0
  Cholesterol (High), Grade 3, n=3: number analyzed (Participants) | 3
  Cholesterol (High), Grade 3, n=3 | 0
  Cholesterol (High), Grade 4, n=3: number analyzed (Participants) | 3
  Cholesterol (High), Grade 4, n=3 | 0
  CPK increased, Grade 0, n=48 | 48
  CPK increased, Grade 1, n=48 | 0
  CPK increased, Grade 2, n=48 | 0
  CPK increased, Grade 3, n=48 | 0
  CPK increased, Grade 4, n=48 | 0
  Creatinine increased, Grade 0, n=48 | 48
  Creatinine increased, Grade 1, n=48 | 0
  Creatinine increased, Grade 2, n=48 | 0
  Creatinine increased, Grade 3, n=48 | 0
  Creatinine increased, Grade 4, n=48 | 0
  Creatinine clearance decreased, Grade 0, n=48 | 39
  Creatinine clearance decreased, Grade 1, n=48 | 0
  Creatinine clearance decreased, Grade 2, n=48 | 9
  Creatinine clearance decreased, Grade 3, n=48 | 0
  Creatinine clearance decreased, Grade 4, n=48 | 0
  Glucose (hyperglycemia), Grade 0, n=48 | 41
  Glucose (hyperglycemia), Grade 1, n=48 | 7
  Glucose (hyperglycemia), Grade 2, n=48 | 0
  Glucose (hyperglycemia), Grade 3, n=48 | 0
  Glucose (hyperglycemia), Grade 4, n=48 | 0
  Glucose (hypoglycemia), Grade 0, n=48 | 48
  Glucose (hypoglycemia), Grade 1, n=48 | 0
  Glucose (hypoglycemia), Grade 2, n=48 | 0
  Glucose (hypoglycemia), Grade 3, n=48 | 0
  Glucose (hypoglycemia), Grade 4, n=48 | 0
  Hypophosphatemia, Grade 0, n=48 | 46
  Hypophosphatemia, Grade 1, n=48 | 2
  Hypophosphatemia, Grade 2, n=48 | 0
  Hypophosphatemia, Grade 3, n=48 | 0
  Hypophosphatemia, Grade 4, n=48 | 0
  Potassium (Hyperkalemia), Grade 0, n=48 | 48
  Potassium (Hyperkalemia), Grade 1, n=48 | 0
  Potassium (Hyperkalemia), Grade 2, n=48 | 0
  Potassium (Hyperkalemia), Grade 3, n=48 | 0
  Potassium (Hyperkalemia), Grade 4, n=48 | 0
  Potassium (Hypokalemia), Grade 0, n=48 | 48
  Potassium (Hypokalemia), Grade 1, n=48 | 0
  Potassium (Hypokalemia), Grade 2, n=48 | 0
  Potassium (Hypokalemia), Grade 3, n=48 | 0
  Potassium (Hypokalemia), Grade 4, n=48 | 0
  Sodium, hypernatremia, Grade 0, n=48 | 48
  Sodium, hypernatremia, Grade 1, n=48 | 0
  Sodium, hypernatremia, Grade 2, n=48 | 0
  Sodium, hypernatremia, Grade 3, n=48 | 0
  Sodium, hypernatremia, Grade 4, n=48 | 0
  Sodium, hyponatremia, Grade 0, n=48 | 48
  Sodium, hyponatremia, Grade 1, n=48 | 0
  Sodium, hyponatremia, Grade 2, n=48 | 0
  Sodium, hyponatremia, Grade 3, n=48 | 0
  Sodium, hyponatremia, Grade 4, n=48 | 0
  Hypertriglyceridemia, Grade 0, n=3: number analyzed (Participants) | 3
  Hypertriglyceridemia, Grade 0, n=3 | 2
  Hypertriglyceridemia, Grade 1, n=3: number analyzed (Participants) | 3
  Hypertriglyceridemia, Grade 1, n=3 | 1
  Hypertriglyceridemia, Grade 2, n=3: number analyzed (Participants) | 3
  Hypertriglyceridemia, Grade 2, n=3 | 0
  Hypertriglyceridemia, Grade 3, n=3: number analyzed (Participants) | 3
  Hypertriglyceridemia, Grade 3, n=3 | 0
  Hypertriglyceridemia, Grade 4, n=3: number analyzed (Participants) | 3
  Hypertriglyceridemia, Grade 4, n=3 | 0
  Uric acid increased, Grade 0, n=48 | 42
  Uric acid increased, Grade 1, n=48 | 6
  Uric acid increased, Grade 2, n=48 | 0
  Uric acid increased, Grade 3, n=48 | 0
  Uric acid increased, Grade 4, n=48 | 0

31. Secondary Outcome: Number of Participants With Maximum Toxicity Post-Baseline in Hematology Parameters: Oral lead-in Phase
Description: Hematology parameters were graded according to DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events as Grade 0: none, Grade 1: mild; Grade 2: moderate; Grade 3: severe; and Grade 4: potentially life-threatening consequences. Higher grade indicates more severity. Clinical hematology parameters included: APTT prolonged, Hb (increased), WBC (decreased), lymphocytes count (decreased), neutrophils (decreased), platelets (decreased), prothrombin international normalized ratio (Pro.INR) (increased). Baseline was the last available assessment prior to the time of the first dose. Maximum toxicity grade reached by a participant post-Baseline was summarized.
Time Frame: Up to Week 4
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB 30 mg (Oral lead-in Phase)
Number analyzed (Participants) | 48
Participants
  APTT prolonged, Grade 0 | 48
  APTT prolonged, Grade 1 | 0
  APTT prolonged, Grade2 | 0
  APTT prolonged, Grade 3 | 0
  APTT prolonged, Grade 4 | 0
  Hb (increased), Grade 0 | 48
  Hb (increased), Grade 1 | 0
  Hb (increased), Grade 2 | 0
  Hb (increased), Grade 3 | 0
  Hb (increased), Grade 4 | 0
  WBC (decreased), Grade 0 | 48
  WBC (decreased), Grade 1 | 0
  WBC (decreased), Grade 2 | 0
  WBC (decreased), Grade 3 | 0
  WBC (decreased), Grade 4 | 0
  Lymphocytes count (decreased), Grade 0 | 48
  Lymphocytes count (decreased), Grade 1 | 0
  Lymphocytes count (decreased), Grade 2 | 0
  Lymphocytes count (decreased), Grade 3 | 0
  Lymphocytes count (decreased), Grade 4 | 0
  Neutrophils (decreased), Grade 0 | 48
  Neutrophils (decreased), Grade 1 | 0
  Neutrophils (decreased), Grade 2 | 0
  Neutrophils (decreased), Grade 3 | 0
  Neutrophils (decreased), Grade 4 | 0
  Platelets (decreased), Grade 0 | 47
  Platelets (decreased), Grade 1 | 1
  Platelets (decreased), Grade 2 | 0
  Platelets (decreased), Grade 3 | 0
  Platelets (decreased), Grade 4 | 0
  Prothrombin INR (increased), Grade 0 | 48
  Prothrombin INR (increased), Grade 1 | 0
  Prothrombin INR (increased), Grade 2 | 0
  Prothrombin INR (increased), Grade 3 | 0
  Prothrombin INR (increased), Grade 4 | 0

32. Secondary Outcome: Number of Participants With Abnormal Urinalysis Parameters: Oral lead-in Phase
Description: as for outcome 4
Time Frame: Up to Week 4
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB 30 mg (Oral lead-in Phase)
Number analyzed (Participants) | 48
Participants
  Protein, Grade 0 | 48
  Protein, Grade 1 | 0
  Protein, Grade 2 | 0
  Protein, Grade 3 | 0
  Protein, Grade 4 | 0

33. Secondary Outcome: Number of Participants With Shift From Baseline in Vital Signs With Respect to Clinical Concern Range: Oral lead-in Phase
Description: Vital signs were measured after participants had rested in supine position for at least 5 minutes. Clinical concern ranges were: SBP (Low <85 mmHg, High: >160 mmHg), DBP (Low: <45 mmHg, High: >100 mmHg), pulse rate (Low: <40 mmHg, High: >100 mmHg). Worst case results are presented. Participants were counted in the worst case category that their value changes to (Low, Normal or High), unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, were recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Time Frame: Up to Week 4
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB 30 mg (Oral lead-in Phase)
Number analyzed (Participants) | 48
Participants
  SBP, To low | 0
  SBP, To Normal or No Change | 48
  SBP, To High | 0
  DBP, To low | 0
  DBP, To Normal or No Change | 48
  DBP, To High | 0
  Pulse rate, To low | 0
  Pulse rate, To Normal or No Change | 48
  Pulse rate, To High | 0

34. Secondary Outcome: Percentage of Participants With Injection Discontinuation-Injection Phase
Description: Percentage of participants with injection discontinuation is presented.
Time Frame: Week 5 to 41
Population: Safety Injection Population
Measure: Number; unit: Percentage of participants
Arm/Group | CAB LA 600 mg (Injection Phase)
Number analyzed (Participants) | 47
Percentage of participants | 4

35. Secondary Outcome: Number of Participants With Grade 2 to 4 Injection Site Pain-Injection Phase
Description: Severity of injection site reactions was analyzed using DAIDS AE Grading Table. The severity is categorized into grades as following: Grade 1 (mild): causing no or minimal interference with usual social and functional activities, Grade 2 (moderate): causing greater than minimal interference with usual social and functional activities, Grade 3 (severe): causing inability to perform usual social and functional activities, Grade 4 (Potentially life threatening): causing inability to perform basic self-care functions or hospitalization indicated. Higher grade indicates more severe condition. Number of participants who had at least one Grade 2 to 4 Injection site reaction is presented.
Time Frame: Week 5 to 41
Population: Safety Injection Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg (Injection Phase)
Number analyzed (Participants) | 47
Participants | 18

36. Secondary Outcome: HIV-Prevention Treatment Satisfaction Total Score-Injection Phase
Description: HIV-Prevention Treatment Satisfaction Questionnaire (change) (HIV-PrevTSQc) was used to assess participant tolerability and satisfaction to the treatment. It consisted total 13 questions. The experience of HIV prevention treatment was assessed using a scale from 3 (much more satisfied/effective/convenient/ flexible/likely to recommend the treatment/likely to speak well of the treatment/easier now) to -3 (much less satisfied/effective/convenient/flexible/likely to recommend the treatment/likely to speak well of the treatment/easier now). Total score was calculated by taking sum of scores of all questions. It ranges from -39 to 39, with higher scores indicating more satisfaction.
Time Frame: At Week 10
Population: Safety Injection Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | CAB LA 600 mg (Injection Phase)
Number analyzed (Participants) | 45
Scores on scale | 23.7 (8.55)

37. Secondary Outcome: Number of Participants With Acceptability of Cabotegravir for HIV Prevention
Description: Number of participants who consider using cabotegravir for HIV prevention in the future is presented. Participants were asked if they would consider using cabotegravir for HIV prevention in the future and their answers to this question were recorded as 'Yes', 'No' or 'Missing'.
Time Frame: Up to Week 41
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir
Number analyzed (Participants) | 48
Participants
  Yes | 40
  No | 7
  Missing | 1

38. Other Pre Specified Outcome: Relationship Between Safety and Tolerability Parameters With Cabotegravir PK Parameters
Description: Relationship between safety and tolerability parameters with cabotegravir PK parameters was planned to be analyzed.
Time Frame: Up to Week 41
Population: Safety Population. This was a conditional secondary endpoint for which results are not available because population pharmacokinetic (Pop PK) analyses were not conducted.
Arm/Group | Cabotegravir
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected up to Week 4 for oral-lead in phase; Weeks 5 to 41 for Injection phase and Weeks 42 to 89 for long-term follow-up phase.
Description: AEs and SAEs were collected in the Safety Population for Oral-lead in, Safety injection Population for Injection Phase and long-term follow up phase.
Groups:
- CAB 30 mg - Oral lead-in Phase: Participants received 30 mg Cabotegravir tablet once daily orally for 4 weeks during oral lead-in phase.
- CAB LA 600 mg - Injection Phase: Participants received CAB LA 600 mg administered as a single 3 mL intramuscular injection on Weeks 5, 9, 17, 25 and 33 during Injection phase.
- CAB LA 600 mg - Long-term Follow-up Phase: After Injection phase, participants were followed-up till Week 89 (long-term follow-up phase).
Arm/Group | CAB 30 mg - Oral lead-in Phase | CAB LA 600 mg - Injection Phase | CAB LA 600 mg - Long-term Follow-up Phase
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/48 | 1/47 | 0/47
Other Adverse Events (participants affected / at risk) | 13/48 | 47/47 | 17/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAB 30 mg - Oral lead-in Phase (N=48) | CAB LA 600 mg - Injection Phase (N=47) | CAB LA 600 mg - Long-term Follow-up Phase (N=47)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAB 30 mg - Oral lead-in Phase (N=48) | CAB LA 600 mg - Injection Phase (N=47) | CAB LA 600 mg - Long-term Follow-up Phase (N=47)
Mouth ulceration (Gastrointestinal disorders) | 3 | 2 | 0
Injection site induration (General disorders) | 0 | 4 | 0
Injection site pain (General disorders) | 0 | 47 | 0
Injection site pruritus (General disorders) | 0 | 3 | 0
Injection site swelling (General disorders) | 0 | 22 | 0
Pyrexia (General disorders) | 0 | 9 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 3
Tonsillitis (Infections and infestations) | 0 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 15 | 9
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 2
Headache (Nervous system disorders) | 1 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2 | 2
Alanine aminotransferase increased (Investigations) | 1 | 2 | 4
Blood uric acid increased (Investigations) | 1 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT03422172/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT03422172/SAP_001.pdf